CLINICAL TRIAL: NCT05450562
Title: A Phase 1/2 Open-label, First-in-human, Dose Escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of SAR444200-based Regimen in Participants With Advanced Solid Tumors.
Brief Title: Dose Escalation and Expansion Study of SAR444200-based Regimen in Adult Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD17240; U1111-1264-3207 (Registry Identifier: ICTRP); 2021-006623-17 (EudraCT Number)
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR444200 - Dose Escalation Phase (Part 1A) (Experimental): SAR444200 will be administered as intravenous injection as monotherapy in participants with GPC3+ solid tumors over a 21-day cycle
  Interventions: Biological: SAR444200
- SAR444200 - Dose Expansion Phase (Part 2A) (Experimental): SAR444200 will be administered as intravenous injection in participants with GPC3+ NSCLC over a 21-day cycle
  Interventions: Biological: SAR444200
- SAR444200 and Atezolizumab combination therapy - Dose Escalation Phase (Part 1B) (Experimental): SAR444200 in combination with atezolizumab will be administered as intravenous injection in participants with GPC3+ solid tumors over a 21-day cycle
  Interventions: Biological: SAR444200; Biological: Atezolizumab

INTERVENTIONS:
Biological: SAR444200 — Sterile lyophilized powder for solution for infusion Route of administration: intravenous (IV) infusion
Biological: Atezolizumab — concentrate for solution for infusion Route of administration: intravenous (IV) infusion
  Other Names: Tecentriq®
  Arms: SAR444200 and Atezolizumab combination therapy - Dose Escalation Phase (Part 1B)

SUMMARY:
This is Phase 1/Phase 2, open label, multiple cohort, first-in-human study to evaluate safety, PK, PDy and efficacy of SAR444200 as a monotherapy or in combination with other anti-cancer agents for participants aged at least 18 years with previously treated metastatic malignancies.

DETAILED DESCRIPTION:
Treatment Period: enrolled participants will receive continuous treatment until disease progression (PD), unacceptable adverse event (AE), or other permanent discontinuation criteria.

The End of Treatment visit will occur 30 days ±7 days from last IMP administration or prior to initiation of further therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis for participants for Part 1A and Part 1B:

  1. Metastatic and/or unresectable HCC diagnosed by histology and/or cytology, or diagnosed clinically by the American Association for the Study of Liver Diseases (AASLD) criteria for participants with liver cirrhosis (participants without liver cirrhosis must be diagnosed histologically) OR Other histology/cytology proven advanced and/or metastatic non-HCC solid tumors
  2. Not amenable to available standard of care: participants must have experienced disease progression on/after standard of care, or no acceptable standard curative or palliative treatments exist (or are no longer effective), according to Investigator judgement, or the participant declines standard of care therapy.
* Cancer diagnosis for participants for Part 2A:

  1. Metastatic NSCLC with no actionable driver gene mutants (such as epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK)), diagnosed by histology and/or cytology not amenable to available standard of care and must have progressed on/after therapy that included an anti-PD(L)-1 agent with or without platinum-based chemotherapy.
  2. Progressive disease should be observed during the course of anti-PD(L)-1 therapy or within 12 weeks from the last dose of anti-PD(L)-1 therapy
* Additional for Part 2A: At least 1 measurable lesion per RECIST 1.1 criteria
* For all participants:

  1. Positive GPC3 expression on tumor tissue as determined locally or centrally
  2. Capable of giving signed informed consent

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥2.
* Predicted life expectancy ≤3 months.
* For participants with HCC: Child Pugh Class B or C liver score within 14 days of initiation of IMP. Participants with Child Pugh Class B-7 score are allowed for Part 1A.
* Known active brain metastases or leptomeningeal metastases.
* History of allogenic or solid organ transplant
* Treatment-related immune-mediated (or immune-related) AEs from immune-modulatory agents (including but not limited to anti-PD1/PD-L1 agents and anti-cytotoxic T lymphocyte associated protein 4 monoclonal antibodies) that caused permanent discontinuation of the agent, or that were Grade 4 in severity
* Significant cardiovascular disease within 3 months prior to initiation of IMP, uncontrolled arrhythmia requiring medication, or unstable angina.
* Ongoing AEs caused by any prior anti-cancer therapy >Grade 2
* Known uncontrolled human immunodeficiency virus (HIV), hepatitis B infection, or known untreated current hepatitis C infection
* Known second malignancy either progressing or requiring active treatment within the last year.
* For combination therapy: Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events
* Receipt of a live-virus vaccination within 28 days of planned treatment start.
* For Part 2A, has received prior GPC3 targeted anticancer treatment.
* Current pneumonitis or interstitial lung disease, or history of interstitial lung disease or pneumonitis that required oral or IV glucocorticoids to assist with management.

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Part 1A and 1B: Number of participants with Dose Limiting Toxicities (DLTs) | For Part 1A: from the Cycle 1, Day 1 up to Day 21For Part 1B: from Cycle 2 Day 1 up to Day 21
  Incidence and nature of DLTs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Part 1A and 1B: Number of participants with Adverse Events (AEs) | the time from the first dose of study interventions up to 30 days after last dose of study interventions
  Incidence of treatment emergent AEs and serious adverse events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Part 2A: Objective Response Rate (ORR) | From baseline to the end of expansion study (up to 2 years)
  ORR defined as the proportion of participants who have a complete response (CR) or partial response (PR) determined per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Part 1A and 1B: Objective Response Rate (ORR) | Baseline to end of dose escalation study (up to 2 years)
  ORR defined as the proportion of participants who have a complete response (CR) or partial response (PR) determined per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
All parts: Duration of response (DoR) | Baseline to end of study (up to 2 years)
  DoR defined as the time from first documented evidence of confirmed CR or PR until progressive disease (PD) or death from any cause, whichever occurs first determined per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
All parts: Assessment of PK parameters: Cmax | Cycle 1 Day 1 to Day 21
  Maximum plasma concentration observed
All parts:Assessment of PK parameters: AUC0-T | Cycle 1 Day 1to Day 21
  Area under the concentration versus time curve calculated using the trapezoidal method during a dosing interval (T)
All parts: Assessment of PK parameters: Tmax | Cycle 1 Day 1to Day 21
  Time to reach Cmax
All parts: Incidence of anti-drug antibodies (ADAs) to SAR444200 | From the first dose of Cycle to 30 days after last dose of study interventions. Cycle duration is 21 days
  Incidence of participants with anti-drug antibodies to SAR444200
All parts: Incidence of anti-drug antibodies (ADAs) to atezolizumab | From the first dose of Cycle to 30 days after last dose of study interventions. Cycle duration is 21 days
Part 2A: Progression Free Survival (PFS) | From baseline to end of expansion study (up to 2 years)
  PFS, defined as the time from the date of first IMP administration to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 (or death due to any cause, whichever occurs first)
Part 2A: Number of participants with Adverse Events (AEs) | The time from the first dose of study interventions up to 30 days after last dose of study interventions.
  Incidence of treatment emergent AEs and serious adverse events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (4):
  - USC Norris Comprehensive Cancer Center- Site Number : 8400004, Los Angeles, California
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400005, New York, New York
  - Lifespan Corporation- Site Number : 8400002, Providence, Rhode Island
  - The University of Texas MD Anderson Cancer Center- Site Number : 8400003, Houston, Texas
- Canada (2):
  - Investigational Site Number : 1240002, Toronto, Ontario
  - Investigational Site Number : 1240001, Québec, Quebec
- China (2):
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560002, Wuhan
- Singapore (3):
  - Investigational Site Number : 7020002, Singapore
  - Investigational Site Number : 7020003, Singapore
  - Investigational Site Number : 7020001, Singapore
- South Korea (2):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TCD17240 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25349&tenant=MT_SNY_9011